CLINICAL TRIAL: NCT00006364
Title: Phase I and Pilot Study of Subcutaneous Homoharringtonine in Chronic Myelogenous Leukemia
Brief Title: Homoharringtonine in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02360; ID 99-032; N01CM17003 (NIH); CDR0000068237 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Homoharringtonine

ARMS (1):
- Treatment (omacetaxine mepesuccinate) (Experimental): Remission induction therapy: Patients receive remission induction therapy comprising homoharringtonine IV continuously over 24 hours on day 1 and then subcutaneously (SC) twice daily on days 2-14 for course 1. Subsequent courses of remission induction therapy comprise homoharringtonine SC twice daily on days 1-14. Treatment continues monthly for at least 2 courses.
  Maintenance therapy: Patients with complete hematologic remission receive maintenance therapy comprising homoharringtonine SC twice daily on days 1-7 monthly for 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: omacetaxine mepesuccinate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: omacetaxine mepesuccinate — Given IV or SC
  Other Names: CGX-635; homoharringtonine
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of homoharringtonine in treating patients who have chronic phase chronic myelogenous leukemia. Drugs used in chemotherapy, such as homoharringtonine, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of homoharringtonine in patients with transformed phases of chronic myelogenous leukemia (CML). (Phase I completed as of 2/11/2004.) II. Determine the toxicity profile of this drug in these patients. III. Determine the response duration in patients with chronic phase CML treated with this drug.

IV. Compare the pharmacokinetics of this drug administered as a continuous infusion vs subcutaneously in these patients.

OUTLINE: This is a pilot, dose-escalation study. (Phase I completed as of 2/11/2004.)

Remission induction therapy: Patients receive remission induction therapy comprising homoharringtonine IV continuously over 24 hours on day 1 and then subcutaneously (SC) twice daily on days 2-14 for course 1. Subsequent courses of remission induction therapy comprise homoharringtonine SC twice daily on days 1-14. Treatment continues monthly for at least 2 courses.

Maintenance therapy: Patients with complete hematologic remission receive maintenance therapy comprising homoharringtonine SC twice daily on days 1-7 monthly for 3 years in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of homoharringtonine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. An additional cohort of 25-30 patients with chronic phase chronic myelogenous leukemia receives remission induction and maintenance therapy as above at the MTD. (Phase I completed as of 2/11/2004.)

Patients are followed every 3 months.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic phase chronic myelogenous leukemia (CML), as defined by the following:

  * Less than 15% blasts in the peripheral blood (PB) or bone marrow (BM)
  * Less than 20% basophils in the PB or BM
  * Platelet count > 100,000/mm^3 (unless related to therapy)
  * Absence of clonal evolution*
* Philadelphia chromosome- OR BCR/ABL-positive disease by cytogenetics, fluorescence in situ hybridization, or polymerase chain reaction
* Failed prior therapy with imatinib mesylate, as defined by any of the following:

  * Failed to achieve or have lost a complete hematologic remission after 3 months of therapy
  * Failed to achieve or have lost at least a minimal cytogenetic response after 6 months of therapy
  * Failed to achieve or have lost a major or complete cytogenetic response after 12 months of therapy
  * Unable to tolerate imatinib mesylate despite adequate dose adjustment
* Failed no more than 2 prior treatment regimens (in addition to imatinib mesylate)

  * Treatment with hydroxyurea is not considered one regimen
* Ineligible for known regimens or protocols of higher efficacy or priority
* Performance status - Zubrod 0-2
* At least 2 months
* Bilirubin no greater than 2.0 mg/dL
* Creatinine less than 2.0 mg/dL
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Fertile patients must use effective contraception

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1999-11; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of homoharringtonine as assessed by the National Cancer Institute (NCI) Common Terminology Criteria (CTC) | 14 days
Complete hematologic remission (CHR) defined as at least 4 weeks of bone marrow (less than 5% blasts) and peripheral blood with WBC < 10 x 10^9/L and no peripheral blasts, promyelocytes, or myelocytes | Up to 6 years
  Using a Bayesian approach.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States